CLINICAL TRIAL: NCT03782415
Title: Phase 1b/2a Single-center, Open-label, Dose Escalation Study to Evaluate the Safety, Tolerability, and Efficacy of MN-166 (Ibudilast) and Temozolomide Combination Treatment in Patients With Newly Diagnosed or Recurrent Glioblastoma
Brief Title: Study to Evaluate Ibudilast and TMZ Combo Treatment in Newly Diagnosed and Recurrent Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MediciNova (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MN-166-GBM-1201
Record Dates: First submitted 2018-12-17; First posted 2018-12-20 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Glioblastoma; Recurrent Glioblastoma; GBM; Newly Diagnosed Glioblastoma
Keywords: MN-166; GBM; glioblastoma; recurrent GBM; temozolomide; newly diagnosed glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — ibudilast; Temozolomide

STUDY DESIGN:
Intervention Model Description: Phase 1b/2a Single-center, Open-label, Dose-escalation study followed by a fixed-dose study to evaluate the safety, tolerability, and preliminary efficacy of MN-166 plus temozolomide in patients with newly diagnosed or recurrent glioblastoma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MN-166 and temozolomide (Experimental): Part 1: Combination treatment of MN-166 60 mg/day (30 mg twice a day) for 28 days and temozolomide 150 mg/m² on Days 1-5 of 28-day cycle. Part 2: Open-label, fixed-dose MN-166 and temozolomide combination treatment for 6 cycles until disease progression, unacceptable tolerability and/or toxicity or loss of life.
  Interventions: Drug: MN-166; Drug: Temozolomide

INTERVENTIONS:
Drug: MN-166 — MN-166 is an anti-inflammatory/neuroprotective agent. MN-166 distributes well to the CNS (Sanftner et al. 2009) and it is a selective inhibitor of certain cyclic nucleotide phosphodiesterases (PDE) and the pro-inflammatory cytokine, macrophage migration inhibitory factor (MIF). At clinically-relevant plasma or CNS concentrations, MN-166 selectively inhibits macrophage migration inhibitory factor (MIF) (Cho et al 2010) and, secondarily, PDE3, 4 and 10 (Gibson et al 2006).
  Other Names: ibudilast
Drug: Temozolomide — Temozolomide is an oral chemotherapy drug. It is an alkylating agent used as a treatment of some brain cancers; and a first-line treatment for glioblastoma multiforme.
  Other Names: TMZ; Temodar; Temodal; Temcad

SUMMARY:
Part 1 is an open-label, single-arm, dose escalation study of MN-166 (ibudilast) and temozolomide (TMZ) combination treatment. Evaluate safety and tolerability of ibudilast (MN-166) and TMZ combination treatment for 1 cycle (28 days); determine dosage in dose-finding study. Part 2 will evaluate efficacy of fixed-dose MN-166 (ibudilast) and TMZ combination treatment for 6 cycles (~6 months) until disease progression, unacceptable tolerability and/or toxicity or loss of life.

DETAILED DESCRIPTION:
This is a single-center open-label, dose-escalation study to evaluate the safety, tolerability and efficacy of MN-166 (ibudilast) and Temozolomide combination treatment in patients with newly diagnosed or recurrent glioblastoma. To be eligible, subjects are histologically confirmed glioblastoma or gliosarcoma, or astrocytomas with molecular features of glioblastoma, WHO Grade 4. Recurrent glioblastoma patients must have a Karnofsky Performance Status (KPS) ≥70 or Eastern Cooperative Oncology Group (ECOG) performance status of 0-2. Patients having newly diagnosed glioblastoma, gliosarcoma, or astrocytomas with molecular features of glioblastoma must have a KPS ≥60 and ECOG score 0-1. This is divided into a dose-escalation phase (Part 1) followed by a fixed-dose phase (Part 2).

Part 1 will evaluate the safety and tolerability of MN-166 when given in combination with temozolomide, and determine the dose of MN-166 to be used in Part 2 of the study. Up to 18 adult subjects are planned to be enrolled in Part 1.

Part 2 will evaluate the efficacy of MN-166 and temozolomide combination treatment as measured by the proportion of subjects who are progression-free at 6 months. Other outcome measures include the evaluation of overall survival, response rate, and median six-month progression-free survival up to 2 years and up to 50 subjects are planned to be enrolled in Part 2.

ELIGIBILITY:
Major Inclusion Criteria for Recurrent GBM Patients:

1. Age 18 or older;
2. Histologically confirmed GBM (glioblastoma), WHO Grade 4;
3. Patients must have a Karnofsky Performance Status (KPS) ≥70 or Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 (see Appendix 7);
4. Previously received standard front-line GBM treatment including maximal surgical resection followed by external beam radiation therapy and TMZ therapy. Prior use of NovoTTF (Optune) and Gliadel wafers is allowed;
5. Patients must be in first relapse;

   1. Relapse is defined as progression following initial therapy (i.e., radiation and/or chemotherapy). The intent therefore is that patients had no more than 1 prior therapy (i.e., initial treatment). If the patient had a surgical resection for relapsed disease and no anti-cancer therapy was instituted for up to 12 weeks, and the patient undergoes another surgical resection, this is considered to constitute one (1) relapse;
   2. Documented recurrence or progression by brain MRI imaging ≤14 days before study registration;
   3. Measurable disease by RANO criteria (≥ 10 mm x 10 mm).

Major Inclusion criteria for newly diagnosed patients:

1. Ages 18 or older;
2. Newly diagnosed glioblastoma or gliosarcoma (WHO Grade 4) confirmed by histology or astrocytomas with molecular features of gliobastoma;
3. Starting maintenance therapy with temozolomide (150 mg/m^2 on Days 1-5 every 28 days) within 4 weeks prior to screening phase;
4. If patient is receiving corticosteroid, dose must be stable or decreasing for at least 5 days prior to the scan. If steroids are added or the steroid dose is increased between the date of the pretreatment MRI and the start of study, a new baseline MRI or CT scan is required;
5. Karnofsky Performance Status ≥60 at time of screening;
6. ECOG score of 0 or 1 at time of screening;
7. Life expectancy of at least 3 months.

Exclusion Criteria (applied to all patients):

1. History of Grade 2 (CTCAE v4.0) or greater intracranial or intratumoral hemorrhage confirmed by either MRI or CT scan;
2. Current use of anticoagulant treatment with coumadin (low-molecular-weight heparin and factor Xa inhibitors are permitted);
3. Any systemic illness or unstable medical condition that might pose additional risk, including: cardiac, unstable metabolic or endocrine disturbances, renal or liver disease;
4. Patients with a history of a different malignancy except the following circumstances:

   1. They have been disease-free for at least 2 years prior to starting study drug and are deemed by the investigator to be at low risk for recurrence of that malignancy. Patients with the following cancers are eligible if diagnosed and treated within the past 2 years: i. Cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin;

7) Patients who have not recovered to ≤ Grade 1 toxicity by NCI CTCAE v4.0 from the toxic effects of previous therapy with exception of lymphopenia, alopecia and fatigue; 9) For use of other investigational drug or other anti-tumor treatment, the following time periods must have elapsed from the projected start of scheduled study treatment:

1. 4 weeks or 5 half-lives (whichever is shorter) from any investigational agent;
2. 4 weeks from cytotoxic therapy (except 23 days for TMZ; 6 weeks from nitrosoureas);
3. 6 weeks from antibodies treatment (i.e., anti-VEGF antibody);
4. 4 weeks or 5 half-lives (whichever is shorter) from other anti-tumor therapies;
5. 2 days from NOVO-TTF (Optune®).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-12-29 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Evaluate safety and tolerability of ibudilast and temozolomide combination treatment | 1-6 months
  Determine the proportion of patients with
  * Treatment-emergent adverse events (TEAEs) as measured by the CTCAE v4.0 and
  * Treatment discontinuations due to TEAEs and Dose-Limiting Toxicities (DLTs).
Evaluate efficacy of ibudilast and TMZ combination treatment | 1-6 months
  Proportion of patients who are progression free at 6 months (PFS6) using the RANO criteria.

SECONDARY OUTCOMES:
Evaluate Tmax | 1-6 months
  Time from start of dosing at which the maximum concentration is observed)
Cmax | 1-6 months
  Maximum observed concentration)
AUC | 1-6 months
  Area under the concentration versus time curve from the start of dose administration to the last quantifiable point within the dosing interval.
Terminal rate constant | 1-6 months
  Calculated from the terminal slope of the log-linear regression of concentration with time.
Terminal half-life | 1-6 months
  Time required for the plasma concentration of a drug to decrease 50% in the final stage of its elimination
Maximum tolerated dose determination | 1-6 months
  Determine maximum tolerable dose of ibudilast taken in combination with TMZ
Evaluate the safety of fixed-dose ibudilast in combination with TMZ | 1-6 months
  Reporting of treatment-emergent adverse events
  * Treatment-emergent adverse events (TEAEs) as measured by the CTCAE v4.0 and
  * Treatment discontinuations due to TEAEs and Dose-Limiting Toxicities (DLTs).
Evaluate overall survival, response rate, and median 6-month progression-free survival (PFS6) | 1-6 months
  Overall survival will be measured for each subject with time origin at the date of Study Day 1 until recorded date or death or last follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Kazuko Matsuda, MD PhD MPH, Study Director — MediciNova, Inc.
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho Y, Crichlow GV, Vermeire JJ, Leng L, Du X, Hodsdon ME, Bucala R, Cappello M, Gross M, Gaeta F, Johnson K, Lolis EJ. Allosteric inhibition of macrophage migration inhibitory factor revealed by ibudilast. Proc Natl Acad Sci U S A. 2010 Jun 22;107(25):11313-8. doi: 10.1073/pnas.1002716107. Epub 2010 Jun 8. PMID 20534506
- [Background] Gibson LC, Hastings SF, McPhee I, Clayton RA, Darroch CE, Mackenzie A, Mackenzie FL, Nagasawa M, Stevens PA, Mackenzie SJ. The inhibitory profile of Ibudilast against the human phosphodiesterase enzyme family. Eur J Pharmacol. 2006 May 24;538(1-3):39-42. doi: 10.1016/j.ejphar.2006.02.053. Epub 2006 Mar 13. PMID 16674936
- [Background] Sanftner LM, Gibbons JA, Gross MI, Suzuki BM, Gaeta FC, Johnson KW. Cross-species comparisons of the pharmacokinetics of ibudilast. Xenobiotica. 2009 Dec;39(12):964-77. doi: 10.3109/00498250903254340. PMID 19925385